CLINICAL TRIAL: NCT05791110
Title: Diagnostic Value of Fecal Pancreatic Elastase 1 in the Diagnosis of Pancreatic Exocrine Insufficiency: a Multi-center Study
Brief Title: PE-1 in the Diagnosis of Pancreatic Exocrine Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PE1-PEI
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Pancreatic Exocrine Insufficiency
Keywords: PE-1; Pancreatic exocrine insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pancreatic exocrine function (Other): Strict clinical diagnosis and fecal pancreatic elastase 1 test were performed for each subject (including PEI patients (n=525) and non-PEI patients (n=528))
  Interventions: Diagnostic Test: Fecal pancreatic elastase 1 test

INTERVENTIONS:
Diagnostic Test: Fecal pancreatic elastase 1 test — Fecal pancreatic elastase 1 test are immunoassays for the quantitative determination of fecal pancreatic elastase in human stool samples.

SUMMARY:
The aim of this study was to evaluate and determine the clinical performance of Fecal Pancreatic Elastase 1 Test in the diagnosis of pancreatic exocrine insufficiency.

DETAILED DESCRIPTION:
Fecal Pancreatic Elastase 1 (PE-1)Test has high diagnostic accuracy in pancreatic exocrine insufficiency (PEI), has become a painless noninvasive diagnostic modality in clinical practice, and has been widely used in clinical practice.

However, in China, the diagnostic ability of the PE-1 test in the Chinese population has not been demonstrated and has not been reported. Meanwhile, pancreatin stimulation, 13C-mixed triglyceride breath test, and N-benzoyl-L-tyrosyl-p-aminobenzoic acid test required drugs, which cannot pass the examination of the drug administration and were not allowed to be carried out to diagnose PEI in China. In addition pancreatin stimulation is an invasive test has certain risks for subjects and 72-hour fecal fat quantification was mainly used for the diagnosis of severe PEI. Therefore, This study adopted strict clinical diagnosis as a comparative method for PE-1 test to judge the ability of PE-1 test to diagnose PEI in the Chinese population.

This study aims to clarify the application efficacy of PE-1 test in PEI through a multi-center, prospective clinical study comparing PE-1 test with strict clinical diagnosis. To study the accuracy of PE-1 test in the diagnosis of PEI.

ELIGIBILITY:
Inclusion Criteria:

- 【patients with clinical diagnosed PEI】

1. Inpatients or outpatients of both sexes, aged 18 to 80 years.
2. Patients with pancreatic disease or after pancreatic or gastric resection (one of the following)

   1. Chronic pancreatitis.
   2. At least 3 months after pancreatectomy (surgical procedures included total pancreatectomy, pancreaticoduodenectomy, pylorus-preserving pancreaticoduodenectomy, and distal pancreatectomy).
   3. Patients recovering from severe acute pancreatitis (duration less than 24 months).
   4. More than 3 months after gastrectomy (surgical methods included total gastrectomy, proximal gastrectomy, and distal gastrectomy).
3. Enrolled patients had at least one of the following symptoms (except those after pancreatectomy)

   1. abdominal distension.
   2. Weight loss (weight loss is defined as loss of more than 5% of basal body weight in one year).
   3. steatorrhea.
4. Agreed to participate in the study and signed an informed consent form.

【patients without clinical diagnosed PEI】

1. Both male and female, aged between 18 and 80 years old.
2. Patients who met one of the following criteria were included in the study:

   1. Patients with functional gastrointestinal diseases who had no history of pancreatectomy, gastrectomy, or abdominal radiotherapy were included.
   2. Healthy volunteers.
   3. Patients with benign hepatobiliary diseases, thyroid, breast diseases, and digestive tract diseases who had no history of pancreatectomy, gastrectomy, or abdominal radiotherapy were included.
3. Agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

1. Pregnant women
2. Critically ill patients
3. The subjects with mental disorders were unable to cooperate with the researchers
4. patients who had undergone ileocolon bladder replacement surgery or complicated with intestinal obstruction and other diseases that could not collect feces
5. the quantity of fecal samples, storage and transportation conditions of samples do not meet the requirements of the kit
6. patients who underwent two or more times of gastrectomy or pancreatectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Reliability of fecal pancreatic elastase 1 test in the diagnosis of PEI | 1 week
  Diagnostic consistency (kappa value) of fecal pancreatic elastase 1 test

SECONDARY OUTCOMES:
Accuracy of fecal pancreatic elastase 1 test in the diagnosis of PEI | 1 week
  Diagnostic sensitivity, specificity, positive likelihood ratio, negative likelihood ratio of fecal pancreatic elastase 1 test
Predictive value of fecal pancreatic elastase 1 test in the diagnosis of PEI | 1 week
  Positive predictive value, negative predictive value of fecal pancreatic elastase 1 test
Accuracy, reliability, and predictive of fecal pancreatic elastase 1 test in the diagnosis of severe PEI | 1 week
  Severe PEI was defined as PE-1 content in feces less than 100μg/g. Diagnostic consistency (kappa value), sensitivity, specificity, positive likelihood ratio, negative likelihood ratio, positive predictive value, negative predictive value of fecal pancreatic elastase 1 test in severe PEI.

CONTACTS AND LOCATIONS:
Overall Officials: zhuan liao, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No